CLINICAL TRIAL: NCT05637138
Title: Influence of Temperature on Transcutaneous Blood Gas Diffusion: CAPNOS Project
Acronym: CAPNOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC22.0188
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers, Pathologies for Which paCO2 Monitoring is Crucial, Particularly in the Context of Chronic Obstructive Pulmonary Disease (COPD)

STUDY DESIGN:
Intervention Model Description: only one group of healthy volunteers is planned in the study, for which measurements of skin permeability, subcutaneous microcirculation and TcpO2 / oxygen sensor will be performed.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Other): The totality of the measurements will be carried out on a single visit following the obtaining of the consent (obtained the same day or during a preceding visit).
  The total duration of this single visit, including the time of information, the collection of consent and all the measurements is estimated at 2 hours per subject.
  Before the installation of the different measuring devices, a preliminary interview and a clinical examination will be carried out in order to verify in particular the absence of skin lesions.
  The measurement of subcutaneous microcirculation (no unit) and tcpO2 (kPa) will be carried out simultaneously with the measurement of CO2 diffusion (main criterion), during a single session of measurements at 5 different temperatures (non-thermostated, then thermostated at 35, 38, 41 and 44°C)
  Interventions: Device: tcpCO2 measure; Device: tcpO2 measure; Device: measurement of tissue conductivity to CO2: KS; Device: measurement of microcirculation

INTERVENTIONS:
Device: tcpCO2 measure — Measurement of tcpCO2 by medical grade sensor: non-thermostatted, at 35°C, 38°C, 41°C and 44°C
Device: tcpO2 measure — Measurement of tcpO2 by medical grade sensor: non-thermostatted, at 35°C, 38°C, 41°C and 44°C
Device: measurement of tissue conductivity to CO2: KS — measurement of tissue conductivity to CO2: KS by CAPNOS sensor : non-thermostatted, at 35°C, 38°C, 41°C and 44°C
Device: measurement of microcirculation — measurement of microcirculation by CAPNOS sensor : non-thermostatted, at 35°C, 38°C, 41°C and 44°C

SUMMARY:
The measurement of tcpCO2 has many disadvantages: the need for regular calibration (4 to 8 hours) of the sensor, the fact that the sensor heats the skin (risk of burns), the impossibility of measurement in ambulatory and the high cost of the monitor. In order to develop a new type of tcpCO2 sensor, it is necessary to acquire knowledge in fundamental physiology on the diffusion of CO2 through the skin.

DETAILED DESCRIPTION:
From a clinical point of view, the arterial carbon dioxide (CO2) pressure - paCO2 - is a particularly interesting physiological data because it gives information on the proper functioning of the cardiorespiratory system. However, the current "gold standard" measurement of this paCO2 requires an arterial puncture, an operation that requires qualified personnel, a rapid analysis of the blood samples collected, and entails risks and discomfort for the patient. In fact, the transcutaneous partial pressure of CO2 - tcpCO2 - is often used as an indirect measure for paCO2, due to its good correlation with the latter. However, current tcpCO2 monitors are bulky, expensive (€10-20k), and possess significant drift resulting in the need to recalibrate the measurement electrode every 4-8 hours. Moreover, these monitors heat the skin to temperatures between 41 and 44°C which can lead to burns, especially when used on infants.

Indeed, an alternative to current tcpCO2 monitors seems highly desirable. In particular, in the face of the rise of wearable electronics, a solution approaching wrist-worn pulse oximeters but for CO2 measurement would be an undeniable asset that cannot be achieved without an overhaul of the tcpCO2 measurement technology.

It is in this global context that the present research is set; to develop a portable tcpCO2 sensor, two main avenues are to be explored. On the one hand, it is necessary to know the modalities of CO2 diffusion through the subcutaneous tissues and the skin towards an external medium (ambient air or sensor). On the other hand, it is necessary to develop a reliable technique to measure CO2 by means of a sensor placed against the skin and this with a minimal drift.

The present research focuses exclusively on the first of these two tracks, i.e. on the phenomenon of CO2 diffusion through the skin. Indeed, the literature on this subject is old and incomplete. In particular, the diffusion rate of CO2 through the skin as a function of skin temperature is not known. However, this variation is of crucial interest for the dimensioning of a tcpCO2 sensor in terms of autonomy. Indeed, the CO2 diffusion rate through the skin has a direct influence on the response time of such a sensor.

The present research is therefore purely exploratory, with the objective of acquiring new knowledge in physiology. It aims to fill the gaps in the literature on the variations of transcutaneous CO2 diffusion rate as a function of temperature, with the long-term objective of developing a new type of tcpCO2 sensor circumventing the constraints of current monitors. The aim is not to develop a new type of tcpCO2 sensor, but to characterize the diffusion rate of CO2 through the skin using a system developed specifically for this study. The measurement system used is an experimental device not intended to be marketed as a medical device. Indeed, it measures a CO2 flow rate and not a partial pressure - partial pressure which is, as a reminder, the quantity of clinical interest.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 and under 80 years of age
* Do not present any contraindication (e.g. skin lesions such as eczema, psoriasis,...) to any of the investigations of the study
* Have given their free, informed and written consent

Exclusion Criteria:

* Subjects under 18 or over 80 years of age
* Skin lesion at any of the measurement sites
* Inability to give written informed consent
* Subjects taking vasodilator treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-08-23 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
CO2 diffusion through skin | Day 0
  Measurement of the conductivity of tissues in CO2: Ks variable, by CAPNOS probe in 5 measures: Non-thermostated, 35, 38, 41 and 44°C

SECONDARY OUTCOMES:
Measurement of the subcutaneous microcirculation | Day 0
  Measurement of subcutaneous microcirculation (without unit) at Non-thermostated, 35°C, 38°C, 41°C and 44°C by laser Doppler probe
Measurement of TcpO2 | Day 0
  TcpO2 measurement (kPa) at Non-thermostated, 35°C, 38°C, 41°C and 44°C by oxygen sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Giroux Metges, Brest, France